CLINICAL TRIAL: NCT01007305
Title: Elective Bilateral Salpingo-oophorectomy Versus Ovarian Conservation: A Pilot Randomized, Controlled Trial
Brief Title: Bilateral Oophorectomy Versus Ovarian Conservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Vanessa L. Jacoby, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BSO 01
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2009-11

CONDITIONS: Oophorectomy; Hysterectomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bilateral salpingo-oophorectomy (Experimental): Removal of both ovaries and fallopian tubes at the time of hysterectomy for benign conditions.
  Interventions: Procedure: Bilateral salpingo-oophorectomy
- Ovarian conservation (Active Comparator): No ovaries or fallopian tubes removed at the time of hysterectomy for benign conditions.
  Interventions: Procedure: Ovarian conservation

INTERVENTIONS:
Procedure: Bilateral salpingo-oophorectomy — Removal of both ovaries and fallopian tubes at the time of hysterectomy
  Arms: Bilateral salpingo-oophorectomy
Procedure: Ovarian conservation — Both ovaries and fallopian tubes not removed at the time of hysterectomy
  Arms: Ovarian conservation

SUMMARY:
This is a pilot study to assess the feasibility of conducting a randomized, blinded, controlled trial of bilateral salpingo-oophorectomy (BSO, removal of the ovaries and fallopian tubes) versus ovarian conservation among premenopausal women age 40 years and greater who plan to undergo hysterectomy for a benign gynecologic condition. Subjects will be randomized to BSO or ovarian conservation concomitant with hysterectomy and remain blinded to group assignment. The primary goal of this pilot is to determine the feasibility of recruiting and retaining study participants in anticipation of conducting a larger, multi-centered trial. However, the investigators will also obtain baseline data and follow-up measures at 6 weeks and 6 months after surgery. Outcomes will be assessed in several domains that the investigators hypothesize may be effected by oophorectomy: cardiovascular health, skeletal health, sexual functioning, and health-related quality-of-life.

ELIGIBILITY:
Inclusion Criteria:

1. Plans to undergo hysterectomy for any non-cancerous gynecologic condition, including symptomatic fibroids, abnormal bleeding, pelvic pain, or pelvic organ prolapse. Hysterectomy may be done abdominally, vaginally or laparoscopically
2. Premenopausal defined as having at least one menses in the 3 months prior to surgery
3. Age > or = 40 years
4. Speaks English or Spanish

Exclusion Criteria:

1. Personal or family history of breast and/or ovarian cancer (at least one first degree relative with a diagnosis of breast or ovarian cancer) or a known BRCA mutation
2. Known or suspected adnexal mass by physical exam or radiologic imaging study
3. Gynecologist recommends BSO for treatment of pelvic pain and/or endometriosis
4. Known history of coronary heart disease defined as any of the following: prior myocardial infarction, history of angioplasty, history of angina, admission to the hospital for evaluation of chest pain, or use of nitroglycerin to treat angina
5. History of stroke
6. History of osteoporosis

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | start of study
Flow-mediated diameter of the brachial artery | Baseline and 6 months follow-up
Serum bone turnover markers | Baseline and 6 months follow-up
Sexual functioning and quality-of-life questionnaires | Baseline and 6 month follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, Sans Francisco, San Francisco, California